CLINICAL TRIAL: NCT03735836
Title: Effect of Fish Oil Monoglycerides on the Omega-3 Index: Pilot Study (IO3-02)
Brief Title: Effect of Fish Oil Monoglycerides on the Omega-3 Index
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Samuel Fortin (Industry)
Responsible Party: Sponsor-Investigator, Samuel Fortin, Principal Investigator, SCF Pharma
Organization: SCF Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IO3-02
Record Dates: First submitted 2018-11-02; First posted 2018-11-08 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Pharmacokinetic in Normal Population

STUDY DESIGN:
Intervention Model Description: Randomized study with two parallel treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MaxSimil 2 capsules daily (Experimental): Subjects will receive two (2) capsules per day of MAG-EPA/MAG-DHA omega-3 oils for a total of 600mg of MAG-EPA and 260mg of MAG-DHA daily during 20 consecutive weeks of treatment.
  Interventions: Other: MAG-EPA/MAG-DHA omega-3 oils
- MaxSimil 3 capsules daily (Experimental): Subjects will receive two (3) capsules per day of of MAG-EPA/MAG-DHA omega-3 oils for a total of 900mg of MAG-EPA and 390mg of MAG-DHA daily during 20 consecutive weeks of treatment.
  Interventions: Other: MAG-EPA/MAG-DHA omega-3 oils

INTERVENTIONS:
Other: MAG-EPA/MAG-DHA omega-3 oils — The monoglyceride (MAG) eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) are chemically modified fish oils that fall into the Natural Health products category in Canada.

SUMMARY:
The objective of this study is to establish the pharmacokinetic curve for two different doses of MaxSimil at steady-state over a 20-week period, namely two (2) or three (3) tablets per day. MaxSimil is a concentrated fish oil monoglyceride (MAG) that facilitates absorption of the omega-3 oils by the body. Each capsule contains 300 mg of monoglyceride eicosapentaenoic acid (MAG-EPA) and 130 mg of monoglyceride docosahexaenoic acid (MAG-DHA). Thirty-two (32) subjects will be enrolled and randomly assigned to one of the two parallel treatment doses. Pharmacokinetics will be assessed by measuring the omega-3 index at eight (8) different times during the study. A first sample will be taken before the start of treatment and then every four (4) weeks during treatment. Then, two last measurements of the omega-3 index will be done at four (4) and seven (7) weeks after the end of treatment. Apart from the study treatment and collection of samples for the measurement of the omega-3 index, the only other interventions will be the measurement of body weight at screening and at the end of the study, pregnancy test for women at screening, questioning for demographic information and for the follow-up of the subject's health and concomitant medication intake.

DETAILED DESCRIPTION:
Thirty-two (32) subjects will be enrolled and randomly assigned to one of the two parallel treatment doses. The study population will be men and women of 19 years and older, with no allergy or history of allergy to fish. Participants must not have taken omega-3 supplements in the last 60 days prior to study enrollment. Pregnant or lactating women will be excluded from the study.

The objective of this study is to establish the pharmacokinetic curve for two different doses of MaxSimil at steady-state over a 20-week period of treatment, namely two (2) or three (3) tablets per day. MaxSimil is a concentrated monoglyceride (MAG) form of omega-3 fish oil that is better absorbed by the body compared to regular fish oil. Each capsule contains 300 mg of monoglyceride eicosapentaenoic acid (MAG-EPA) and 130 mg of monoglyceride docosahexaenoic acid (MAG-DHA).

Pharmacokinetics will be assessed by measuring the omega-3 index at eight (8) different times during the study. A first blood sample will be taken before the start of treatment and then at week four (4), eight (8), twelve (12), sixteen (16) and twenty (20). Then, two last measurements of the omega-3 index will be done at four (4) and seven (7) weeks after the end of treatment. The samples will all be taken by capillary puncture during visits at the clinic. A total of nine (9) visits may be done including the recruitment/screening/enrollment visit. Visit 1 could be done immediately after enrollment for a total of eight (8) visits instead of nine.

The screening tasks include pregnancy testing for women, measurement of the omega-3 index, body weight and height, recording of the baseline health status and concomitant treatment. Then, for visits 2 to 5, study treatment will be dispensed, returned and accounted, blood sample will be collected for the measurement of the omega-3 index, and the health status will be followed for any adverse event outcome.

Visits 6 to 8 are post-treatment follow-ups where omega-3 index testing will be done as well as the follow-up of the health status and concomitant medication intake.

ELIGIBILITY:
Inclusion Criteria:

1. Participant of at least 19 years old.
2. Available for the entire duration of the study and willing to participate based on the information provided in the informed consent form (ICF) duly read and signed by the latter.
3. Absence of intellectual problems likely to limit the validity of consent to participate in the study or the compliance with protocol requirements, ability to cooperate adequately, to understand and observe the instructions of the coordinator of the study.
4. Participant having no difficulty swallowing tablets or capsules.

Exclusion Criteria:

1. Known allergy to fish or history of allergic reactions attributable to fish, or a compound similar to fish oil.
2. Females who are pregnant or lactating, or has tested positive to a pregnancy test at screening.
3. Participant who used omega-3 supplements within 60 days prior to Day 1 of the study.
4. Participant who, in the opinion of the research coordinator, may not be able to comply with the requirements of the protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Measurement of the Omega-3 index over time to establish the Pharmacokinetic curve and bioavailability at steady state. | 12 months
  The objective of this pilot study is to collect preliminary bioavailability data for two different daily doses of MaxSimil at steady-state, that to say 600mg/260mg and 900mg/490mg daily of EPA/DHA. Blood samples will be taken by capillary puncture at specific time points during treatment and will be analysed to establish the omega-3 index (the fraction of EPA + DHA in the total fatty acids contained in red blood cells) which serves as bioavailability marker.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Clinique Gestion Santé de la Baie, Maria, Quebec
  - Clinique GSM du Littoral, Pointe-au-Père, Quebec

IPD SHARING:
Plan to Share IPD: No